CLINICAL TRIAL: NCT02526693
Title: RAPDx Pupillography for Early Detection of Glaucoma
Brief Title: Is the RAPDx Pupillograph Able to Distinguish Between Glaucoma Subjects and Healthy Subjects?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, George L. Spaeth MD, Principal Investigator, Wills Eye
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-400E
Record Dates: First submitted 2015-08-06; First posted 2015-08-18 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Glaucoma
Keywords: glaucoma; relative afferent pupillary defect; pupillography
MeSH Terms: conditions — Glaucoma; Pupil Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glaucoma Patients (Other): Glaucoma patients recruited from Wills Eye Hospital Glaucoma Service will be tested with the relative afferent pupillary defect test (RAPDx) Pupillometer. The noninvasive RAPDx measures the pupils response during light stimulation.
  Interventions: Diagnostic Test: Pupillometer
- Healthy Controls (Other): Healthy subjects with no eye diseases recruited from Wills Eye Hospital Glaucoma Service staff, family and friends will be tested with the relative afferent pupillary defect test (RAPDx) Pupillometer. The noninvasive RAPDx measures the pupils response during light stimulation.
  Interventions: Diagnostic Test: Pupillometer

INTERVENTIONS:
Diagnostic Test: Pupillometer — The Konan RAPDx (relative afferent pupillary defect) (Konan Medical USA, Irvine, CA) pupillometer utilizes digital, high-definition, infrared machine-vision with eye-tracking and automated blink detection technology to analyze and quantify pupillary response to light.
  Other Names: Relative afferent pupillary defect pupillometer

SUMMARY:
The Konan RAPDx (Konan Medical USA, Irvine, CA) is a newly patented pupillography device.The aims of this study are to assess the ability of the RAPDx to distinguish between healthy subjects and patients with confirmed glaucoma using standard testing sequences developed for use at the Wills Eye Hospital Glaucoma Research Center and to determine the combination of demographic, clinical, and RAPDx testing parameters which allow for maximum sensitivity and specificity.

DETAILED DESCRIPTION:
The RAPDx utilizes noninvasive digital, high-definition, infrared machine-vision with eye-tracking and automated blink detection technology to analyze and quantify the pupillary response to light.

During the scheduled appointment, all patients will receive an undilated fundus examination by the attending ophthalmologist. The following data will be collected; Demographic information, Visual acuity, Intraocular pressure (IOP) measured by Goldmann applanation tonometry, Disc damage likelihood scale (DDLS), Vertical cup/disc ratio, Gonioscopy (if not documented in the chart within the past 2 years) and Humphrey visual field examination.

Each participant will undergo RAPDx testing with two different testing sequences. They are separated by a 10-second resting period during which the patient is instructed to close his or her eyes. The exam may be paused at any time and re-alignment may be performed during any pause. The two testing sequences are:

1. Standard Factory Setting: 0.1-second stimuli with 2-second inter-stimuli pauses;
2. Custom Setting: 3-second stimuli with 1-second inter-stimuli pauses

ELIGIBILITY:
Inclusion Criteria:

Glaucoma patients:

* optic nerve damage (neuroretinal rim notch, asymmetric inter-eye cup to disc (c/d_ ratio >0.2 or disc damage likelihood scale (DDLS) >2, or absence of neuroretinal rim not due to other cause)
* glaucomatous visual field (VF) deficits (cluster of 3 or more points on pattern deviation plot depressed below 5% level, at least 1 depressed below 1% level; OR corrected pattern standard deviation/pattern standard deviation significant at P <0.05; or glaucoma hemifield test "outside normal limits") with good reliability indices (fixation losses, false-positive rate, false-negative rate each < 33%).

Healthy subjects:

* normal optic nerve exam
* normal reliable VF (Humphrey mean deviation (MD) >-2 or Octopus MD ≤0.8; fixation losses, false-positive rate, and false-negative rate each < 33%)
* open angles gonioscopy.

Exclusion Criteria:

* Abnormal ocular motility preventing binocular fixation (e.g. strabismus, nystagmus).
* Any condition preventing adequate visualization and examination of pupil or optic nerve (e.g. dense corneal opacities or lens opacities).
* Active infection of anterior or posterior segments of the eye.
* Any intraocular surgical or laser procedure within previous 4 weeks.
* Any non-glaucomatous condition causing RAPD, anisocoria or corectopia (ex. optic neuropathy, Horner's syndrome, previous iris injury due to trauma or surgery, etc.).
* Subjects under age 18 or subjects presently housed in correctional facility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Spaeth, MD, Principal Investigator — Wills Eye Hospital

IPD SHARING:
Plan to Share IPD: No
Manuscript is has not been finalized.

RESULTS

PARTICIPANT FLOW:
Groups:
- Glaucoma Patients: 50 Glaucoma patients recruited from Wills Eye Hospital Glaucoma Service will be tested with RAPDx Pupillometer machine.
  RAPDx Pupillometer: Konan relative afferent pupillary defect RAPDx (Konan Medical USA, Irvine, CA) utilizes digital, high-definition, infrared machine-vision with eye-tracking and automated blink detection technology to analyze and quantify pupillary response to light.
- Healthy Controls: 50 Healthy subjects with no eye diseases from Wills Eye Hospital Glaucoma Service staff, family and friends will be tested with RAPDx Pupillometer machine.
  RAPDx Pupillometer: Konan relative afferent pupillary defect RAPDx (Konan Medical USA, Irvine, CA) utilizes digital, high-definition, infrared machine-vision with eye-tracking and automated blink detection technology to analyze and quantify pupillary response to light.
Period: Overall Study
Arm/Group | Glaucoma Patients | Healthy Controls
Started | 53 | 51
Completed | 50 | 50
Not Completed | 3 | 1
Not completed — Physician Decision | 3 | 1

BASELINE CHARACTERISTICS:
Population: 4 participants enrolled were excluded from analysis due to other comorbidities or abnormal values of measurement parameters. Three excluded participants were from the Glaucoma Group, one was from the Control Group.
Groups:
- Glaucoma: Glaucoma patients are recruited from Wills Eye Hospital glaucoma service, who will be tested with the RAPDx Pupillography machine.
  RAPDx Pupillography: The Konan RAPDx (Konan Medical USA, Irvine, CA) utilizes digital, high-definition, infrared machine-vision with eye-tracking and automated blink detection technology to analyze and quantify the pupillary response to light.
- Healthy Control: Healthy subjects are recruited from Wills Eye Hospital primary care service, who will be tested with the RAPDx Pupillography machine.
  RAPDx Pupillography: The Konan RAPDx (Konan Medical USA, Irvine, CA) utilizes digital, high-definition, infrared machine-vision with eye-tracking and automated blink detection technology to analyze and quantify the pupillary response to light.
- Total: Total of all reporting groups
Arm/Group | Glaucoma | Healthy Control | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 34 | 57
  >=65 years | 27 | 16 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 19 | 17 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 37 | 14 | 51
  White | 9 | 29 | 38
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Glaucoma patients were recruited from Wills Eye Hospital Glaucoma Service, Philadelphia, PA, USA. Healthy controls were recruited from staff, friends and family members of Wills Eye Hospital Glaucoma Research Center.
  participants
    United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Amplitude Asymmetry of Pupil Constriction
Description: Pupil size changes when light shines into the eyes making the diameter of the pupil smaller (constriction). The size of the pupil's reaction to light, measured in millimeters, is the amplitude or change in diameter. Amplitude of maximum pupil constriction (pupil size) when light is shone is compared between the right and left eyes. Asymmetry is the difference between maximum pupil size of the two eyes.
Time Frame: 1 examination, one hour
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Glaucoma Patients: Glaucoma patients recruited from Glaucoma Service at Wills Eye Hospital will be tested with RAPDx Pupillography machine
  Relative afferent pupillary defect RAPDx Pupillography: The Konan RAPDx (Konan Medical USA, Irvine, CA) utilizes digital, high-definition, infrared with eye-tracking and automated blink detection to analyze and quantify pupillary response to light and dark with a standard testing sequence and a custom sequence.
- Healthy Controls: Healthy subjects are recruited from the Wills Eye clinic, who will be tested with the RAPDx Pupillography machine
  Relative afferent pupillary defect RAPDx Pupillography: The Konan RAPDx (Konan Medical USA, Irvine, CA) utilizes digital, high-definition, infrared with eye-tracking and automated blink detection to analyze and quantify pupillary response to light and dark with a standard testing sequence and a custom sequence.
Arm/Group | Glaucoma Patients | Healthy Controls
Number analyzed (Participants) | 50 | 50
millimeters
  Custom sequence | 0.8 (0.75) | 0.29 (0.27)
  Standard sequence | 0.5 (0.52) | 0.16 (0.12)

2. Primary Outcome: Latency Asymmetry of Pupil Constriction
Description: Pupil size changes at different speeds when light shines into the eyes making the diameter of the pupil smaller (constriction). The speed of the pupil's reaction to light is the latency or amount of time. Latency of maximum pupil constriction when light is shone is compared between the right and left eyes. Asymmetry is the difference in time it takes for maximum pupil constriction between the two eyes.
Time Frame: 1 examination, one hour
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Glaucoma: 50 Glaucoma patients recruited from Wills Eye Hospital Glaucoma Service will be tested with RAPDx Pupillometer.
  RAPDx Pupillometer: The Konan relative afferent pupillary defect RAPDx (Konan Medical USA, Irvine, CA) utilizes digital, high-definition, infrared machine-vision with eye-tracking and automated blink detection technology to analyze and quantify pupillary response to light and dark with a standard testing sequence and a custom sequence.
- Healthy Controls: 50 Healthy subjects with no eye diseases recruited from Wills Eye Hospital Glaucoma Service staff, family and friends will be tested with the relative afferent pupillary defect test (RAPDx) Pupillometer.
  Pupillometer: The Konan RAPDx (relative afferent pupillary defect) (Konan Medical USA, Irvine, CA) pupillometer utilizes digital, high-definition, infrared machine-vision with eye-tracking and automated blink detection technology to analyze and quantify pupillary response to light and dark with a standard testing sequence and a custom sequence.
Arm/Group | Glaucoma | Healthy Controls
Number analyzed (Participants) | 50 | 50
milliseconds
  Custom sequence | 0.22 (0.23) | 0.14 (0.14)
  Standard sequence | 0.2 (0.21) | 0.13 (0.11)

3. Primary Outcome: Maximum Constriction Asymmetry Duration
Description: Log difference between duration of maximum pupil constriction when light is shone into the right versus the left eye. The duration of maximum constriction is calculated as time in milliseconds between point of maximum constriction and time when pupil amplitude has reached 50% of peak amplitude of dilation.
Time Frame: 1 examination, one hour
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Glaucoma Patients: 50 Glaucoma patients recruited from Wills Eye Hospital Glaucoma Service will be tested with relative afferent pupillary defect (RAPDx) Pupillometer.
  Pupillometer: The Konan RAPDx (relative afferent pupillary defect) (Konan Medical USA, Irvine, CA) pupillometer utilizes digital, high-definition, infrared machine-vision with eye-tracking and automated blink detection technology to analyze and quantify pupillary response to light and dark with a standard testing sequence and a custom sequence.
- Healthy Controls: 50 Healthy subjects with no eye diseases recruited from Wills Eye Hospital Glaucoma Service staff, family and friends will be tested with relative afferent pupillary defect (RAPDx) Pupillometer.
  Pupillometer: The Konan RAPDx (relative afferent pupillary defect) (Konan Medical USA, Irvine, CA) pupillometer utilizes digital, high-definition, infrared machine-vision with eye-tracking and automated blink detection technology to analyze and quantify pupillary response to light and dark with a standard testing sequence and a custom sequence.
Arm/Group | Glaucoma Patients | Healthy Controls
Number analyzed (Participants) | 50 | 50
milliseconds | 2.23 (0.64) | 1.92 (0.54)

ADVERSE EVENTS:
Time Frame: 1 examination, one hour
Groups:
- Glaucoma Patients: 50 Glaucoma patients recruited from Wills Eye Hospital Glaucoma Service were tested with RAPDx Pupillometer.
  Konan (Konan Medical USA, Irvine, CA) RAPDx (relative afferent pupillary defect) test utilizes digital, high-definition, infrared machine-vision with eye-tracking and automated blink detection technology to analyze and quantify pupillary response to light.
- Healthy Controls: 50 Healthy controls recruited from Wills Eye Hospital Glaucoma Service staff, family and friends were tested with RAPDx Pupillometer.
  Konan (Konan Medical USA, Irvine, CA) RAPDx (relative afferent pupillary defect) test utilizes digital, high-definition, infrared machine-vision with eye-tracking and automated blink detection technology to analyze and quantify pupillary response to light.
Arm/Group | Glaucoma Patients | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
Small sample size. Single site design. Single light design limits pupil stimulus.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No